CLINICAL TRIAL: NCT01929772
Title: German Lactat Clearance in Severe Sepsis
Acronym: GLASS
Status: Completed | Type: Observational
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Other Study IDs: 12-052
Record Dates: First submitted 2013-08-19; First posted 2013-08-28 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Severe Sepsis; Septic Shock
MeSH Terms: conditions — Sepsis; Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- severe sepsis or septic shock: patients with severe sepsis or septic shock

SUMMARY:
The aim of this study is to investigate if there is a correlation between lactate clearance and the course at patients with severe sepsis and septic shock at german intensive care units.

ELIGIBILITY:
Inclusion Criteria:

* Patients with severe sepsis or septic shock
* signed informed consent

Exclusion Criteria:

* severe sepsis or septic schock within 4 weeks before inclusion of study
* shock of other genesis
* persons being accomondated in an institution because of court or official order
* persons being interdependet to the investigator
* employees of the investigator

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with severe sepsis or septic shock
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2012-09; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Lactate Clearance | Within 6 hours after diagnoses
  Determination of lactate clearance within 6 hours after diagnosis of severe sepisis and septic shocik

SECONDARY OUTCOMES:
SOFA Score | Day of hospitalization, day 7, day 8

OTHER OUTCOMES:
Mortality | After 28 days
  Determination of the mortality of the collective after 28 days
Duration intensive care unit and hospitalization | 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- Department for Operative Intensive Care and Intermediate Care - University Hospital Aachen, Aachen, North Rhine Westfalia, Germany